CLINICAL TRIAL: NCT04987879
Title: NASH AMPK Exercise Dosing (AMPED) Trial
Acronym: AMPED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Christopher Sciamanna, MD, MPH, Professor, Department of Medicine and Public Health Sciences, Penn State Health Milton S Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00018280; K23DK131290 (NIH)
Record Dates: First submitted 2021-07-13; First posted 2021-08-03 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-07

CONDITIONS: NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Exercise Arm 1 (Experimental): Aerobic exercise will be completed by walking, jogging or running or by using cardio equipment (e.g., recumbent bike). Each session will begin with a warm-up with walking and dynamic exercises. A 5-min walking cool down will end the session. The training dose for this arm is 750 MET-min/wk for 3-5 days per week, 22-45 minutes per session at a moderate to vigorous intensity. The exercise can be completed in person or virtually.
  Interventions: Behavioral: Exercise
- Exercise Arm 2 (Experimental): Aerobic exercise will be completed by walking, jogging or running or by using cardio equipment (e.g., recumbent bike). Each session will begin with a warm-up with walking and dynamic exercises. A 5-min walking cool down will end the session. The training dose for this arm is 1,000 MET-min/wk for 3-5 days per week, 30-60 minutes per session at a moderate to vigorous intensity. The exercise can be completed in person or virtually.
  Interventions: Behavioral: Exercise
- Standard of Care (No Intervention): This group will receive best NASH clinical practices counseling at baseline and end-of-trial in accordance with NAFLD clinical practice guidelines and be reinforced by handouts from the American Liver Foundation.

INTERVENTIONS:
Behavioral: Exercise — Aerobic exercise can be completed by walking, jogging or running or by using cardio equipment (e.g., recumbent bike). Each session will begin with a warm-up with walking (30-40% target HR for 5-min) and dynamic exercises (knee-to-chest, 10-yd lateral shuffle, bent over twist, calf sweeps, leg swings). A 5-min walking cool down will end the session (30-40% target HR).
  Other Names: Physical activity
  Arms: Exercise Arm 1; Exercise Arm 2

SUMMARY:
There is no known cure or regulatory agency approved drug therapy for nonalcoholic fatty liver disease (NAFLD), the leading cause of liver disease worldwide, and its progressive type, NASH. This places increased importance on using exercise to treat NAFLD.

While physical activity is recommended for all with NAFLD, how to best prescribe exercise as a specific treatment remains unknown, including what dose of exercise is most effective.

DETAILED DESCRIPTION:
The mechanism explaining how exercise training benefits patients with NAFLD and NASH is unclear. The AMPK pathway may be responsible for the benefits seen with exercise training because: 1) AMPK has a liver-specific role in hepatic de novo lipogenesis and fatty acid oxidation, 2) AMPK activity is abnormally low in NAFLD and 3) NAFLD animal models demonstrate exercise changes the liver-specific AMPK pathway, leading to less liver fat accumulation by reducing lipogenesis and increasing fatty acid oxidation (This has not been studied in patients). Importantly, exercise-induced AMPK activation appears to be dose dependent.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-69 years
* Sedentary [<90 min/wk of exercise identified by the Get Active Questionnaire (GAQ)
* BMI >25kg/m2
* Liver biopsy within six months prior to enrollment showing:

  * NASH defined by NASH Clinical Research Network (CRN) histology scoring system (NAS) >4 and MRI-PDFF >5% and;
  * Liver fibrosis stage 1-3

Exclusion Criteria:

* Active cardiac symptoms
* Body mass index (BMI) >45kg/m2
* Cancer that is active
* Inability to walk >2 blocks
* Institutionalized/prisoner
* Other liver disease
* Pregnancy
* Secondary hepatic steatosis
* Severe comorbidities
* AUDIT-C questionnaire identified significant alcohol use
* Substance abuse/active smoking
* Uncontrolled diabetes (changes in drug dosing over previous three months or A1c >9%)
* GAQ response indicates exercise may be unsafe.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-08-30 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Change in liver fat | 16 weeks
  Degree of liver fat change as measured by magnetic resonance imaging proton density fat fraction (MRI-PDFF) across different doses of exercise in patients with NASH.

SECONDARY OUTCOMES:
Hip/waist circumference | 16 weeks
  change in Hip/waist circumference
Body mass index | 16 weeks
  change in body mass index
change in body composition | 16 weeks
  change in body composition as measured by Dual-energy X-ray absorptiometry (DXA scan) across different doses of exercise in patients with NASH.
Insulin | 16 weeks
  change in insulin
Hemoglobin A1c | 16 weeks
  change in Hemoglobin A1c
change in cholesterol and triglycerides levels (dyslipidemia) | 16 weeks
  change in cholesterol and triglycerides levels (dyslipidemia) as measured by clinical labs.
Interleukin-6 | 16 weeks
  change in Interleukin-6
c-reactive protein | 16 weeks
  change in c-reactive protein
Non-Alcoholic Fatty Liver Disease (NAFLD) Fibrosis Score | 16 weeks
  change in NAFLD Fibrosis Score which estimates amount of scarring in the liver based on several laboratory tests.
  NAFLD Score Correlated Fibrosis Severity < -1.455 F0-F2
  -1.455 - 0.675 Indeterminant score > 0.675 F3-F4 Fibrosis Severity Scale
  F0 = no fibrosis F1 = mild fibrosis F2 = moderate fibrosis F3 = severe fibrosis F4 = cirrhosis
Enhance liver fibrosis (ELF) test | 16 weeks
  change in Enhance liver fibrosis (ELF) test
TIMP-1 | 16 weeks
  change in TIMP-1
ProC3 | 16 weeks
  change in ProC3
Adiponectin | 16 weeks
  change in Adiponectin
Fibroblast Growth Factor (FGF) 21 | 16 weeks
  change in Fibroblast Growth Factor (FGF) 21
Change in stiffness of the liver | 16 weeks
  Change in stiffness of the liver as measured by the technique of transient elastography, a non-invasive test to stage the severity of liver disease.
Liver glycogen | 16 weeks
  change in liver glycogen

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Sciamanna, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No